CLINICAL TRIAL: NCT00030576
Title: A Phase I/II Study Of OSI-774 In Combination With Cisplatin In Patients With Recurrent Or Metastatic Squamous Cell Cancer Of The Head And Neck
Brief Title: Erlotinib and Cisplatin in Treating Patients With Recurrent or Metastatic Head and Neck Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000069178 (PHL-002); PMH-PHL-002; NCI-5380; CAN-NCIC-IND157
Record Dates: First submitted 2002-02-14; First posted 2003-01-27 (Estimated); Last update posted 2018-10-10 (Actual); Status verified 2018-10

CONDITIONS: Head and Neck Cancer
Keywords: recurrent metastatic squamous neck cancer occult primary; neck cancer with occult primary squamous carcinoma; stage IV squamous cell carcinoma of the lip and oral cavity; recurrent squamous cell carcinoma of the lip and oral cavity; stage IV squamous cell carcinoma of the oropharynx; recurrent squamous cell carcinoma of the oropharynx; stage IV squamous cell carcinoma of the nasopharynx; recurrent squamous cell carcinoma of the nasopharynx; stage IV squamous cell carcinoma of the hypopharynx; recurrent squamous cell carcinoma of the hypopharynx; stage IV squamous cell carcinoma of the larynx; recurrent squamous cell carcinoma of the larynx; squamous cell carcinoma of paranasal sinus and nasal cavity; recurrent squamous cell carcinoma of sinus and nasal cavity
MeSH Terms: conditions — Head and Neck Neoplasms; Squamous Cell Carcinoma of Head and Neck | interventions — Cisplatin; Erlotinib Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- OSI-774 and cisplatin (Experimental): HNSCC patients treated in three escalating dose cohorts of daily continous oral erlotinib (OSI-774) and intermittent IV cisplatin given every 21 days
  Interventions: Drug: cisplatin; Drug: erlotinib hydrochloride

INTERVENTIONS:
Drug: cisplatin
Drug: erlotinib hydrochloride

SUMMARY:
RATIONALE: Biological therapies such as erlotinib may interfere with the growth of tumor cells and slow the growth of the tumor. Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining erlotinib with cisplatin may kill more tumor cells.

PURPOSE: Phase I/II trial to study the effectiveness of combining erlotinib and cisplatin in treating patients who have recurrent or metastatic head and neck cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the objective response rate in patients with recurrent or metastatic squamous cell cancer of the head and neck treated with erlotinib and cisplatin.
* Determine the stable disease rates, duration of response, progression-free survival, median survival, and overall survival of patients treated with this regimen.
* Determine the safety and tolerability of this regimen in these patients.
* Determine the relationship between clinical, pharmacokinetic, and pharmacodynamic effects of this regimen in these patients.
* Correlate baseline and post-treatment levels of epidermal growth factor receptor, its downstream signaling components, and markers of angiogenesis and apoptosis in tumor and skin biopsies with clinical outcome in patients treated with this regimen.

OUTLINE: This is a dose-escalation, multicenter study.

Patients receive oral erlotinib once daily on days -6 to 21 for the first course only and cisplatin IV over 60 minutes on day 1. For the second and subsequent courses, patients receive oral erlotinib once daily on days 1-21 and cisplatin as in course 1. Treatment repeats every 21 days for up to 6 courses in the absence of disease progression or unacceptable toxicity. Patients with stable or responding disease after 6 courses may continue to receive erlotinib alone until disease progression.

Cohorts of 3-6 patients receive escalating doses of erlotinib and cisplatin until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity. At least 6 patients are treated at the MTD.

Patients are followed every 3 months.

PROJECTED ACCRUAL: A maximum of 43 patients will be accrued for this study within 18 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed squamous cell carcinoma of the head and neck

  * All primary sites, including oral cavity, oropharynx, nasopharynx, hypopharynx, larynx, and paranasal sinus
* Recurrent, unresectable, and/or metastatic disease
* At least 1 measurable lesion

  * At least 20 mm with conventional techniques OR at least 10 mm with spiral CT scan
* Lesions accessible for biopsy
* Tumor specimen available for evaluation of epidermal growth factor receptor (EGFR) expression
* No known brain metastases

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* ECOG 0-2 OR
* Karnofsky 60-100%

Life expectancy:

* More than 12 weeks

Hematopoietic:

* WBC at least 3,000/mm^3
* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3

Hepatic:

* Bilirubin no greater than 1.25 times upper limit of normal (ULN)
* AST and ALT no greater than 2.5 times ULN

Renal:

* Creatinine normal OR
* Creatinine clearance at least 60 mL/min

Cardiovascular:

* No symptomatic congestive heart failure
* No unstable angina pectoris
* No cardiac arrhythmia

Gastrointestinal:

* No gastrointestinal tract disease resulting in malabsorption
* No requirement for IV alimentation
* No active peptic ulcer disease
* Inability to swallow tablets or silicon-based G-tubes allowed

Ophthalmic:

* No abnormalities of the cornea based on history (e.g., dry eye syndrome or Sjogren's syndrome)
* No congenital abnormality (e.g., Fuch's dystrophy)
* No abnormal slit-lamp examination using a vital dye (e.g., fluorescein or Bengal-Rose)
* No abnormal corneal sensitivity test (e.g., Schirmer test or similar tear production test)

Other:

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No other malignancy within the past 5 years except carcinoma in situ of the cervix, nonmelanoma skin cancer, or second primary squamous cell cancer originating from the head and neck
* No grade 2 or greater residual ototoxicity or neuropathy from prior platinum-based therapy
* No significant traumatic injury within the past 21 days
* No other concurrent uncontrolled illness
* No ongoing or active infection
* No psychiatric illness or social situation that would preclude study participation

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* No prior chemotherapy for recurrent or metastatic disease
* Prior platinum-based chemotherapy with radiotherapy or platinum-based induction chemotherapy allowed
* At least 6 months since prior chemotherapy

Endocrine therapy:

* Not specified

Radiotherapy:

* See Chemotherapy
* At least 4 weeks since prior radiotherapy (except low-dose, limited-fraction palliative non-myelosuppressive radiotherapy [e.g., involving less than 20% of functioning bone marrow using 800 cGy in 1 fraction or 2,000 cGy in 5 fractions]) and recovered
* No prior radiotherapy to target lesion unless there is evidence of disease progression

Surgery:

* See Disease Characteristics
* At least 21 days since prior major surgery
* No prior surgical procedure affecting gastrointestinal absorption

Other:

* No prior EGFR-targeting therapies
* No prior investigational agents for recurrent or metastatic disease
* No concurrent combination anti-retroviral therapy for HIV infection
* No other concurrent investigational agents
* No other concurrent anticancer treatment

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2001-11 (Actual); Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lillian L. Siu, MD, FRCPC, Study Chair — Princess Margaret Hospital, Canada; Elizabeth A. Eisenhauer, MD, Study Chair — Cancer Research Institute at Queen's University
Locations (6):
- Canada (6):
  - Margaret and Charles Juravinski Cancer Centre, Hamilton, Ontario
  - Queen's University, Kingston, Ontario
  - Cancer Care Ontario-London Regional Cancer Centre, London, Ontario
  - Ottawa Regional Cancer Centre, Ottawa, Ontario
  - Princess Margaret Hospital, Toronto, Ontario
  - Centre Hospitalier de l'Universite de Montreal, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Agulnik M, da Cunha Santos G, Hedley D, Nicklee T, Dos Reis PP, Ho J, Pond GR, Chen H, Chen S, Shyr Y, Winquist E, Soulieres D, Chen EX, Squire JA, Marrano P, Kamel-Reid S, Dancey J, Siu LL, Tsao MS. Predictive and pharmacodynamic biomarker studies in tumor and skin tissue samples of patients with recurrent or metastatic squamous cell carcinoma of the head and neck treated with erlotinib. J Clin Oncol. 2007 Jun 1;25(16):2184-90. doi: 10.1200/JCO.2006.07.6554. PMID 17538163
- [Result] Siu LL, Soulieres D, Chen EX, Pond GR, Chin SF, Francis P, Harvey L, Klein M, Zhang W, Dancey J, Eisenhauer EA, Winquist E; Princess Margaret Hospital Phase II Consortium; National Cancer Institute of Canada Clinical Trials Group Study. Phase I/II trial of erlotinib and cisplatin in patients with recurrent or metastatic squamous cell carcinoma of the head and neck: a Princess Margaret Hospital phase II consortium and National Cancer Institute of Canada Clinical Trials Group Study. J Clin Oncol. 2007 Jun 1;25(16):2178-83. doi: 10.1200/JCO.2006.07.6547. PMID 17538162
- [Result] Winquist E, Soulieres D, Chen E, et al.: A phase II study of erlotinib in combination with cisplatin in patients with recurrent or metastatic squamous cell cancer of the head and neck (PHL002es/NCIC CTG IND.157). [Abstract] Eur J Cancer 2 (Suppl 8): A-408, 122, 2004.
- [Result] Siu LL, Chen X, Tsao M: A phase I/II study of erlotinib (Tarceva) in combination with cisplatin in patients with recurrent or metastatic squamous cell cancer of the head and neck (HNSCC). [Abstract] Clin Cancer Res 9 (16): A-A92, 2003.